CLINICAL TRIAL: NCT00981812
Title: Clinical Utility and Initial Experience With PEM Flex Solo II PET Scanner and Stereo Navigator Biopsy Accessory for the Diagnosis of Breast Cancer
Brief Title: Positron Emission Mammography (PEM) Biopsy Accessory for the Diagnosis of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Mary Mahoney, Professor, Director of Breast Imaging, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cincinnati-01
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: PET; PEM; Positron Emission Mammography; Breast Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEM Breast Biopsy (Experimental): All patients underwent PEM biopsy.
  Interventions: Procedure: PEM Breast Biopsy

INTERVENTIONS:
Procedure: PEM Breast Biopsy — Breast biopsy using PEM guidance and Stereo Navigator software
  Other Names: Naviscan PEM 2400 Pet Scanner; Stereo Navigator Accessory

SUMMARY:
The purpose of this research study is to evaluate how well the Stereo Navigator Biopsy Accessory for the PEM Flex solo II PET Scanner works for performing breast biopsy on suspicious lesions. This study will also allow the doctors to describe the features of PEM detected lesions and the results obtained using the PEM guided biopsy and will compare the time it took to complete a pre-operative work up using PEM versus MRI in patients with a suspicious breast lesion resulting in cancer.

DETAILED DESCRIPTION:
See brief summary.

ELIGIBILITY:
Inclusion Criteria:

* female
* subject is 25-100 years of age
* subjects has at least one breast imaging finding on mammography and/or ultrasound which is assessed as highly suggestive of malignancy and recommended to biopsy
* subject is able to provide informed consent

Exclusion Criteria:

* subject is pregnant
* subject is actively lactating or discontinued breastfeeding less than 2 months ago
* subject has breast implants
* subject is scheduled for sentinel node procedure using radioactive Tc-99m within 24 hours of the PEM study
* subject has contraindications for core biopsy and other invasive procedures
* subject has Type I diabetes mellitus or poorly controlled Type II diabetes mellitus
* subject has had surgery or radiation therapy on the study breast or has had chemotherapy within the past 12 months
* subject has not fasted for 4-6 hours prior to the procedure and/or have a fasting blood glucose level greater than 140 mg/dl on day of PEM imaging

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Mahoney, MD, Principal Investigator — Univeristy of Cincinnati; Amy Argus, MD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Hospital, The Barrett Center, Cincinnnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from 02/2010 to 06/2011 from University of Cincinnati Medical Center, Radiology Department, Breast Imaging.
Period: Overall Study
Arm/Group | PEM Breast Biopsy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Women 25 or older
Groups:
- Primary: Women 25 years or older with a highly suspicious finding for possible breast cancer on mammography and/or ultrasound, who are to be scheduled for percutaneous breast biopsy.
Arm/Group | Primary
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants] — Women 25 years of age or older with a highly suspicious breast mass recommended to biopsy.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 17
    >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility That Breast Biopsy Can be Performed Using PEM and Stereo Navigator Software After Diagnostic PEM on the Same Day.
Time Frame: At time of biopsy
Measure: Number; unit: Breast Lesions
Groups:
- Lesions Visualized Using Positron Emission Mammography (PEM): Total lesions visualized using positron emission mammography.
Arm/Group | Lesions Visualized Using Positron Emission Mammography (PEM)
Number analyzed (Participants) | 20
Breast Lesions
  Index Lesioins | 22
  Index Lesions Visualized at PEM | 21
  Additional Lesions seen only at PEM | 6
  Lesions technically adequate for targeting | 26
  Number of Lesions Biopsied | 24

ADVERSE EVENTS:
Time Frame: One year and four months.
Arm/Group | PEM Breast Biopsy
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No